CLINICAL TRIAL: NCT04412382
Title: Covid-19: Possible Role of Neutrophil Extracellular Traps
Acronym: NETSINCOVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Chiara Mozzini, Principal Investigator, Azienda Ospedaliera Universitaria Integrata Verona
Other Study IDs: NETS IN COVID-19
Record Dates: First submitted 2020-05-26; First posted 2020-06-02 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Covid-19
Keywords: Covid-19; neutrophil extracellular traps
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- covid-19: Study population: Covid-19 patients aged ≥ 18 years admitted to the Covid sections of the Verona University Hospital. Based on the ongoing epidemic emergency and the lack of specific therapy, we believe that to date this should be the only INCLUSION CRITERION.
  Interventions: Diagnostic Test: NETosis markers
- control: Control group: medical doctors and nurses working in the University Hospital of Verona without known autoimmune diseases nor cancer.
  Interventions: Diagnostic Test: NETosis markers

INTERVENTIONS:
Diagnostic Test: NETosis markers — NETosis markers (Cf-DNA. MPO-DNA, Cit-H3) and the cytokines IL-6 and IL-1β will be analyzed from the subjects' plasma.
  Spittle sample (or bronchoalveolar fluid if necessary for diagnostic-therapeutic purposes) will be collected and the detection of NETs at electron microscopy will be assessed.

SUMMARY:
The process by which neutrophils expel DNA together with various proteins to the outside, forming a network structure called Neutrophil Extracellular Traps (NETs) constitutes a particular cell death that involves the destruction of the nuclear membrane before the plasmatic one. This process is called NETosis and differs from other known forms of cell death, such as necrosis and apoptosis.

This process, however, if exaggerated, brings local or systemic damage. Viruses are known for their ability to evade the body's immune response. Only recently has it been seen that they can act as triggers for NETosis process.

In fact, many viruses can stimulate neutrophils to produce NETs. Virus-induced NETs can begin to circulate in an uncontrolled manner, leading to an extreme systemic response of the body with the production of immunocomplexes, cytokines, Interferon I etc.

To date, there are no data in the literature on the role of NETs in Covid-19 infection, a viral infection that leads to highly lethal interstitial pneumonia and for which there is currently no vaccine or specific therapy.

Advanced forms of Covid-19 are often characterized by hyperinflammation ("cytokine storm") with the development of an ARDS-like condition. Furthermore, reports of micro and macro thrombotic phenomena such as microangiopathy, pulmonary embolism (which has led to a careful evaluation procedure for antithrombotic prophylaxis and/or coagulation in Covid-19 patients) are increasingly frequent.

The primary objective of the study is to understand if NETs can be implicated in the response to Covid-19 and by which mechanisms. Concrete therapeutic proposals could derive from the knowledge and enhancement of this form of innate immunity.

To do this, it will be necessary to evaluate the activity of NETosis in Covid-19 patients and evaluate whether the clinical course of the disease (worsening vs healing) determines the degree of NETosis activity. Therefore, the association between mortality from Covid-19/survival and NETs activity will be studied.

Secondary objectives concern the possibility of studying the associations among NETosis markers and blood inflammation markers and among NETosis markers and the onset of peripheral or deep vein thrombosis.

Finally, the possibility that the plasma deriving from Covid-19 patients could trigger the NETosis process in vitro will be evaluated.

DETAILED DESCRIPTION:
The process by which neutrophils expel DNA together with various proteins to the outside, forming a network structure called Neutrophil Extracellular Traps (NETs) constitutes a particular cell death that involves the destruction of the nuclear membrane before the plasmatic one. This process is called NETosis and differs from other known forms of cell death, such as necrosis and apoptosis.

Neutrophil death by NETs ejection (NETosis) was first described in 2004 by Brinkman.

NETs,as indicated by the word itself, represent a sort of network composed of DNA fibers, histones and proteins derived from the neutrophil granules, whose main function is to trap pathogens (mainly bacteria and fungi).This process is related to the innate immunity.

However, this process, if activated in an exaggerated way, implies itself local or systemic damage.

The DNA expelled during this process is a double stranded DNA, a dsDNA subtype. The dsDNA, which represents a fraction of the DNA available in the circulation (cell free DNA - cfDNA), originates from various processes of cell death, and is therefore correlated with the degree of tissue damage. It is present only in small quantities in healthy subjects.

It is important to underline how during the NETosis process the cellular redox state is altered, leading to an excess production of oxygen free radicals (Reactive Oxygen Species, ROS) and to the activation of the enzyme NADPH oxidase. The formation of NETs, and therefore the process of NETosis, were initially studied in the context of bacterial infections, but subsequently their role became increasingly clear in other conditions such as cancer, autoimmune diseases, lung diseases, atherosclerosis and venous thromboembolic disease.

In particular, NETosis seems to play an important role in all conditions characterized by venous and arterial thrombosis, as numerous evidences have confirmed.

NETosis has also been documented at the microvascular level, such as in vasculitis, thrombotic microangiopathies such as Moschowitz syndrome.

Viruses are known for their ability to evade the body's immune response. Recently it has been seen that they too can act as triggers of NETosis processes.

In fact, many viruses can stimulate neutrophils to produce NETs. Different responses of neutrophils have been seen, from classical NETosis, to the production of antiviral agents or even to the switch to apoptosis.

Virus-induced NETs (therefore complexes of dsDNA, histones, granular proteins) can begin to circulate in an uncontrolled way, leading to an extreme systemic response of the body with the production of immune complexes, cytokines, Interferon I etc.

NETosis appears to be closely linked to the inflammatory response. For example, it is known that in the neutrophilic granulocyte the PAD4 protein is present in the nucleus, it decondensates the chromatin and favors the formation of the NETs. On the other hand, NETs increase in patients with acute respiratory distress syndrome (ARDS) as observed in studies about bronchoalveolar lavage fluid, as well as in patients with acute respiratory failure during COPD exacerbation.

It is therefore clear that virus-induced NETosis acts as a double-edged sword: if on one hand there is the mechanical entrapment of the virus, on the other the inflammatory and immunological reaction triggered by the release of the NETs can be harmful itself.

To date, there are few data in the literature on the role of NETs in Covid-19 infection, a viral infection that can lead to highly lethal interstitial pneumonia and for which there is no vaccine or specific therapy today. Advanced forms of Covid-19 are often characterized by hyperinflammation ("cytokine storm") with the development of an ARDS-like condition. Furthermore, reports of micro and macro thrombotic phenomena such as microangiopathy, pulmonary embolism (which has led to a careful evaluation procedure for antithrombotic prophylaxis and / or coagulation in Covid-19 patients) are increasingly frequent.

OBJECTIVE OF THE STUDY The primary objective of the study is to understand if NETs can be implicated in the response to Covid-19 and by which mechanisms. Concrete therapeutic proposals could derive from the knowledge and enhancement of this form of innate immunity.

To do this, it will be necessary to evaluate the activity of NETosis in Covid-19 patients and evaluate whether the clinical course of the disease (worsening vs healing) determines the degree of NETosi activity. Therefore, the association between mortality from Covid-19/survival and NETs activity will be studied.

Secondary objectives concern the possibility of studying the various associations among NETosis markers and biohumoral indices of inflammation and among NETosi markers and the onset of peripheral or deep vein thrombosis.

Finally, the possibility that the plasma from Covid-19 patients could trigger the NETosis process in vitro will be evaluated.

PLANNED PROCEDURES and COLLECTED INFORMATION Medical examination: (blood pressure, heart rate and SpO2, which will allow to evaluate the precise PaO2 / FiO2 ratio).

As in normal clinical practice, Covid-19 patients will undergo venous sampling for the determination of blood count, creatinine, lipid profile, PCR, D-dimer, LDH, liver function indices and blood glucose.

Precise medical history will be drawn up for each subject. Patients will undergo:electrocardiogram and chest x-ray and, in selected cases, chest CT scan, depending on their clinical need.

They will also undergo venous echo-color Doppler lower limbs examination. A complete analysis of the venous axes will not be necessary. NETosis markers (Cf-DNA. MPO-DNA, Cit-H3) and the cytokines IL-6 and IL-1β will be analyzed from the subjects' plasma.

Spittle sample (or bronchoalveolar fluid if necessary for diagnostic-therapeutic purposes) will be collected and the detection of NETs at electron microscopy will be assessed.

Informed consent will be requested.

CALCULATION OF THE SAMPLE The sample size was defined on the basis of the number of admissions for Covid-19 in the months of March-April 2020 and on the decrease in numbers in the current period.

100 subjects (50 patients and 50 controls) are expected to be enrolled.

STATISTICAL ANALYSIS Hypothetical statistical analysis: the data will be collected through descriptive statistics. The estimates will be accompanied by appropriate 95% confidence intervals. The level of statistical significance is set at 5%. The statistical program Stata 14.2 will be used. Planned test: t-test and Mann-Whitney test. Correlations will be evaluated through Pearson or Spearman coefficients. Furthermore, Kaplan-Meier analyzes will be carried out with the use of Log-Rank test and Cox regression for survival analysis.

ELIGIBILITY:
* Covid-19 patients aged ≥ 18 years admitted to the Covid sections of the Verona University Hospital.
* Control group: medical doctors and nurses working in the University Hospital of Verona.

Exclusion Criteria:

* age <18 years;
* pregnancy;
* known autoimmune diseases.

For the control group:

- positivity to Covid-19 swabs and / or the presence of IgM and IgG antibodies (sierological picture known from the samples taken by the Health surveillance System of the hospital).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population: Covid-19 patients aged ≥ 18 years admitted to the Covid sections of the Verona University Hospital.
  Control group: medical doctors and nurses worìking in the University Hospital of Verona.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
NETOSIS AND MORTALITY | 1 year
  correlation among plasma levels of NETosis markers and Covid-19 mortality
NETOSIS AND DCOVID-19 SEVERITY | 1 year
  correlation among plasma levels of NETosis markers and disease severity (that is duration of hospitalization in days and any need for passage to intensive care with non-invasive ventilation or intubation);

SECONDARY OUTCOMES:
NETOSIS AND INFLAMMATION | 1 year
  correlation among plasma levels of NETosis markers and clinical inflammation biomarkers (white blood cells, PCR IL-6-IL-1β)
NETOSIS AND VENOUS THROMBOSIS | 1 year
  correlation among plasma levels of NETosis markers and the onset of deep vein thrombosis and / or the increase in D-dimer values.

CONTACTS AND LOCATIONS:
Overall Officials: DOMENICO GIRELLI, MD-PhD, Study Chair — Universita di Verona
Locations (1):
- Univeristy of Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: Yes
study protocol and results
Supporting Information: Study Protocol, SAP
Time Frame: end 2020
Access Criteria: mail contact

REFERENCES:
- [Background] Mozzini C, Girelli D. The role of Neutrophil Extracellular Traps in Covid-19: Only an hypothesis or a potential new field of research? Thromb Res. 2020 Jul;191:26-27. doi: 10.1016/j.thromres.2020.04.031. Epub 2020 Apr 27. No abstract available. PMID 32360977